CLINICAL TRIAL: NCT05756829
Title: Type 1 Diabetes Virtual Self-management Education and Support
Acronym: T1ME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Gillian Booth, Nominated Principal Investigator, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTO Project ID: 3644
Record Dates: First submitted 2023-02-09; First posted 2023-03-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High frequency, low-touch virtual health care (Experimental): Participants in this arm will receive a high frequency, low-touch virtual health care intervention through the Maple application, as an adjunct to usual T1D care. High-frequency visits will occur every 2 +/- 1 weeks for a total of 6 months.
  Participants will also receive access to a virtual library to support T1D self-learning and as a guided educational tool.
  Interventions: Other: High frequency, low touch virtual health care
- Standard Care (No Intervention): Participants in this arm will receive the standard of care offered for their condition and by their clinic.

INTERVENTIONS:
Other: High frequency, low touch virtual health care — Virtual visits between certified diabetes educators and patients occurring every 2 +/- 1 weeks for a total of 6 months
  Arms: High frequency, low-touch virtual health care

SUMMARY:
OVERVIEW: People living with type 1 diabetes (T1D) are expected to fit self-management and regular clinical consultations into busy lives. T1D self-management programs that offer frequent contact with care teams are most effective in helping patients achieve optimal glycemic control. However, this is difficult to deliver in the context of current T1D care which involves time-consuming in-person visits during working hours. The proposed study will test a virtual health care intervention to deliver "high frequency, low touch" care aimed at improving metabolic control, while reducing the burden on individuals and their healthcare teams.

STUDY DESIGN: A pragmatic multicenter, open-label, randomized trial to evaluate the short-term effectiveness of a multifaceted virtual health care intervention in improving glycemic control in individuals with T1D. Planned recruitment is 580 participants from 10 specialized T1D centres in Ontario.

INTERVENTION: Our intervention will include 1) frequent, brief virtual visits between patients with T1D and certified diabetes educators (conducted in real time using a secure telemedicine video interface accessible from any PC, tablet or smart phone) combined with automatic appointment reminders, and 2) a centralized web-based platform to provide educational classes, tools, and resources for diabetes self-management. Virtual visits will be an adjunct to routine in-clinic visits for blood pressure monitoring, foot checks, and surveillance for other complications of diabetes. This approach aims to enable patients to receive more education and support than is feasible in traditional health care models, and in a way that is more seamless (i.e. results in fewer disruptions to their daily life) and tailored to their individual needs based on their stage in life.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients ≥18 years of age
2. Physician diagnosis of type 1 diabetes
3. Currently on an insulin pump or using multiple daily insulin injections.
4. HbA1c ≥ 7.5% on most recent laboratory report or estimated from CGM/FGM* report, within the last 4 months

   *14 day look back window, with a wear rate of 70%, based on Estimated A1c or Glucose management Indicator (GMI)
5. Has access to a mobile device or computer/tablet with a video camera
6. Seen for at least one visit in the previous 6 months by participating certified diabetes educator at the selected diabetes clinic OR If a transitioning patient: Currently enrolled in a diabetes program below AND had at least one visit or touch-point prior in the previous 6 months by participating certified diabetes educator at on of our participating diabetes clinics
7. OHIP coverage
8. Currently using an active email address or be willing to obtain an email address
9. Has consistent and reliable access to internet
10. Willing and able to comply with scheduled in-person and virtual visits for 6 month intervention period

Exclusion Criteria:

1. Diagnosed with non-Type 1 diabetes
2. Unable to use a computer/tablet or mobile phone
3. Pregnant
4. On dialysis
5. Unable to fluently speak or read English (self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline HbA1c at 6 months | Baseline, pre-intervention AND Up to 4 weeks after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Booth, MD, Principal Investigator — Unity Health Toronto
Locations (9):
- Canada (9):
  - Waterloo Regional Health Network, Kitchener, Ontario
  - Mackenzie Health, Richmond Hill, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Unity Health Toronto, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Charles H. Best Diabetes Centre, Whitby, Ontario